CLINICAL TRIAL: NCT00162539
Title: Relation Between Maternal Iodine Status and Prenatal Foetal Thyroid Dimension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Christiophe Aucan, Department Clinical Research of Develeppement
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Foetus iodine Status
Record Dates: First submitted 2005-09-10; First posted 2005-09-13 (Estimated); Last update posted 2012-07-26 (Estimated); Status verified 2005-05

CONDITIONS: Deficiency Disease
Keywords: foetal thyroid mensuration
MeSH Terms: conditions — Deficiency Diseases | interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: echography — Correlation of neonatal thyroid volume with maternal iodine deficiency

SUMMARY:
Mother with severe Iodine deficiency are more likely to have neonates with further poor mental development . In order to select population which could benefit from iodine supplementation, ioduria has been tested but cannot be routinely practised. Strong background data suggest that iodine status could be antenatally correlated with foetal thyroid volume. The aim of that study is to examine correlation between these two parameter in a population of 130 healthy pregnant women.

DETAILED DESCRIPTION:
Iodine is an essential element in thyroid homeostasis, particularly in pregnant woman and her fetus. Various studies have clearly shown that antenatal thyroid disorders at both the mother and the fetus could cause in extreme situations of neurological consequences.

At a broader scale, subtle alterations of thyroid hormone balance has been implicated in developmental delays and deviations of the IQ bell curve in newborn infants of mothers with elevated TSH.

The clinical implications of these basic data and public health are yet to confirm.

It has been clearly established that there is a moderate iodine deficiency in France with a decreasing gradient from west to east. In the Ile de France, there is a moderate iodine deficiency, this has led some teams to propose a systematic supplementation of all women in iodine.

One way to target women who really need supplements systematic determination of urinary iodine tongue; this assay is reliable but is difficult to implement in an ad hoc practice at the individual level.

Our team has expertise in the field of fetal thyroid, particularly in its sonographic and reference curves of the perimeter and diameter of the thyroid are now clearly established reliably.

Knowing that iodine deficiency is causing a decline in maternal urine iodine with a phenomenon goitrigénèse and biological hypothyroidism and that some studies have shown that neonatal thyroid volumes were higher in iodine deficient mothers . We postulate that the measurement of fetal thyroid by our criteria can be correlated with maternal urinary iodine.

If this were the case, we will have a simple test to identify iodine supplementation in pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* normal single pregnancy in a healthy volunteer

Exclusion Criteria:

* any associated disease
* pertubation of thyroid status at 12 GA

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2005-10; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
establish a relationship between maternal urinary iodine and thyroid measurements of fetal | final time frame at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Dominique LUTON, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hospital Beaujon, Paris, France

REFERENCES:
- [Derived] Luton D, Alberti C, Vuillard E, Ducarme G, Oury JF, Guibourdenche J. Iodine deficiency in northern Paris area: impact on fetal thyroid mensuration. PLoS One. 2011 Feb 16;6(2):e14707. doi: 10.1371/journal.pone.0014707. PMID 21359193